CLINICAL TRIAL: NCT02225158
Title: Longitudinal Study of Immune Responses to Mycobacterium Tuberculosis (Mtb) in Subjects With Latent Tuberculosis (TB) Infection(LTBI) With or Without Concomitant Helminth Infection
Brief Title: Immune Responses to Mycobacterium Tuberculosis (Mtb) in People With Latent Tuberculosis Infection With or Without Concomitant Helminth Infection
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140178; 14-I-0178
Record Dates: First submitted 2014-08-23; First posted 2014-08-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-05-11

CONDITIONS: Latent Tuberculosis Infection
Keywords: Immunity; Co-Infection; Parasite; Mycobacteria
MeSH Terms: conditions — Latent Tuberculosis; Coinfection; Mycobacterium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

Tuberculosis (TB) is a severe disease and a major cause of death in many people worldwide. It is caused by a bacteria that enters through the lungs and can spread elsewhere in the body. People with latent TB have the bacteria that lie dormant but can become active and cause disease. These people are offered treatment to prevent development of active TB. Worldwide, a lot of people with LTBI also have a parasitic worm called a helminth that can stay in the gut or the blood. These parasites can affect the immune system and cause diseases like TB to become worse. Researchers want to see how helminth infection makes it harder for people to fight TB infection.

Objectives:

- To study how the immune system of people with latent tuberculosis infection (LTBI) acts to prevent development of active TB. Also, to study how helminth infection might affect this immune response.

Eligibility:

* Adults age 18 70 with LTBI as defined by an approved blood test called QuantiFERON TB Gold.
* No evidence of infections like Hepatitis or HIV
* Pregnant subjects and subjects taking medications that suppress the immune system are not eligible.
* Have not received prior treatment for LTBI. Participants might be still eligible if prior treatment for active TB has been received

Design:

Screening phase:

- Participants will be screened with medical history, physical exam, and blood tests for other infections/conditions which might affect the immune system. They will have testing for active TB i.e. blood testing as well as testing of their spit, scans and X-rays.

Baseline phase:

* Only eligible participants will be entered into the study.
* Participants will have interviews, medical history, and physical exam.
* Blood will be drawn from an arm vein for testing.
* Participants will collect stool samples at home for 3 days in a row to test for helminth infection..
* Participants may have apheresis. Blood cells are removed by needle. They pass through a separator machine which returns everything but the cells back to the participant.
* Participants may have procedures at the start and end of the study that let researchers look into the lungs and collect cells.

Study phase, about 2 years:

* All participants will be offered treatment for LTBI which lasts 6-9 months.
* Participants being treated for LTBI will have about 11 study visits. They will visit monthly for 9 months while on treatment, then 6 and 12 months after treatment.
* Participants not eligible/refusing treatment for LTBI will be made aware of active TB, then have 3 other visits, about 6, 12, and 24 months after the baseline visit.
* Participants who have helminth infection will receive appropriate treatment.
* All participants will have blood drawn at each visit.

DETAILED DESCRIPTION:
Mycobacterium tuberculosis (Mtb) infection remains an important cause of morbidity and mortality worldwide. A problem for eradication efforts is the large reservoir of ~2 billion people with latent tuberculosis (TB) infection (LTBI) and poor understanding of factors leading to active disease progression. Helminth infections geographically overlap with Mtb and induce significant immune-mediated modulation. Although CD4+T cells producing IFN-gamma and TNF-alpha have been implicated in protective immunity to TB, a detailed description of the evolution of protective and immunomodulatory responses in LTBI is lacking. Additionally, there is incomplete understanding of how the immunomodulation caused by helminth co-infection affects such responses.

This protocol will attempt to fill this knowledge gap through comprehensive longitudinal immunological analyses of two populations of subjects with LTBI, with or without concurrent helminth infection (HEL+ and HEL- respectively). In both groups, venipuncture and possibly apheresis will be performed to understand protective and modulatory T cell and monocyte/macrophage responses. Subjects will receive treatment for helminth infection and treatment for LTBI will be offered according to current standard of care guidelines. Two groups of subjects within the LTBI group will be offered bronchoscopy and lavage --- (a) those with structural lung damage from prior treated/healed tuberculosis and (b) those with recent prolonged exposure (greater than or equal to 3 months) to a household contact with active TB.

The primary objective is to evaluate CD4+ T cell responses and regulatory T cell responses in HEL+ and HEL- subjects with LTBI at the time of diagnosis (baseline). HEL+ subjects will then receive treatment for parasitic infection and both groups (HEL+ and HEL-) will be offered LTBI treatment. Evolution of the baseline TB-specific immune responses on and after LTBI treatment will then be studied. Additionally, baseline immune responses to mycobacteria will be contrasted in the HEL+ group with all time points post treatment for helminth infection. A secondary objective is to evaluate the immune phenotype and functionality of tissue resident immune cells obtained by bronchoalveolar lavage in subjects with LTBI and structural lung damage from prior treated/healed pulmonary tuberculosis as well as subjects with recent prolonged TB exposure from an active TB case irrespective of helminth infection status.

An exploratory objective is to evaluate if there are subsets of subjects within the LTBI group (irrespective of helminth infection status) who have stable pool of long lasting antigen-specific IL-2 only producing CD4+ central memory T cells and changes to this pool after receiving LTBI treatment.

ELIGIBILITY:
* INCLUSION CRITERIA

All subjects must meet the following criteria:

* Subjects must have 1 of the following:

  * Untreated LTBI, defined as positive Quantiferon TB Gold assay; absence of active TB disease as determined by history, physical examination, chest X-ray, and negative sputum smear and culture for Mtb; and no history of prior treatment for LTBI. OR
  * Chronic inactive TB, defined as past history of documented or selfreported active pulmonary TB for which treatment was received; current negative sputum smear and culture for Mtb; and a positive result on the Quantiferon TB Gold assay. These subjects will compose the treatment-induced LTBI group and will not require treatment for LTBI.
* Age 18-70 years. Subjects over the age of 70 will not be included due to the increased potential for immune senescence
* With or without clinical/microbiologic/serologic evidence of untreated concurrent helminth infection
* Agree to have blood specimens stored for future studies

Subjects undergoing optional bronchoscopy and bronchoalveolar lavage must meet the following additional inclusion criteria:

* Subjects must have 1 of the following:

  * Documented or self reported history of prior treated TB with positive Quantiferon TB Gold test and structural lung findings of chronic inactive tuberculosis on radiologic imaging, defined as: a) calcified Ghon focus with or without apical calcified nodules (Simon foci), b) parenchymal or pleural calcification, and/or c) apical fibrosis and cavitary changes. OR
  * History of recent prolonged (greater than or equal to 3 months) exposure to a confirmed case of active TB disease.
* Able and willing to arrange to have another person drive them home after the procedure
* Able and willing not to eat or drink anything for 6 hours prior and 2 hours after the procedure
* Agree to have respiratory tract samples stored for future research

EXCLUSION CRITERIA

A subject will be excluded if they meet any of the following criteria:

* Presence of active TB disease
* Treatment for helminth infection within the past year
* Positive at screening for HIV, hepatitis B, and/or hepatitis C Cardiovascular instability (Blood pressure: Systolic >180 or <90 mm/Hg or Diastolic >100 or < 50 mm/Hg; pulse <40 or >110)
* Inadequate peripheral venous access
* Anemia (hemoglobin <11 g/dL)
* Current use of corticosteroids or other immunosuppressive agents or documented diagnosis of a primary immunodeficiency disorder
* Underlying heart disease, lung disease, bleeding disorder, or other conditions that, in the judgment of the investigator, contraindicates apheresis
* Temperature greater than or equal to 38.5 degrees C or other clinical evidence of an acute infection at screening
* Currently pregnant or breastfeeding

A subject will not be eligible for optional bronchoscopy and bronchoalveolar lavage if they meet any of the following additional exclusion criteria:

* History of recent/acute clinically significant pulmonary compromise. This will be defined by the following criteria:

  * New lung infection or change in status of chronic lung infection or significant new findings on chest X-ray or CT scan
  * Asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past two years, or that required the use of oral or parenteral corticosteroids during the past two years
  * Clinically significant reactive airway disease that does not respond to bronchodilators
  * Unstable chronic lung disease such as Chronic Obstructive Pulmonary Disease (COPD) or pulmonary fibrosis
  * History of pulmonary hypertension
  * Requirement of supplemental oxygen at rest
* Unstable angina or uncontrolled heart failure or rhythm disturbance
* Significant kidney or liver disease
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions), significant bruising or bleeding difficulties with IM injections or blood draws, or use of anticoagulant medications
* Use of platelet inhibitors including aspirin and NSAIDs within 7 days of procedure or clopidogrel (Plavix [TM]) within 14 days of procedure or the inability to safely stop platelet inhibitors for 7-14 days prior to procedures
* History of allergic reaction to lidocaine, sedative medications like Valium(TM) or Versed (TM), or narcotic medications like morphine or fentanyl
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to bronchoscopy and bronchoalveolar lavage or impairs a volunteer s ability to give informed consent for the procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-08-15; Primary Completion 2017-05-11 (Actual); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
Define the immunologic differences in CD4+ T cell responses between helminth-infected and uninfected subjects with concomitant latent TB at the time of diagnosis and on serial follow-up. | Pre Treatment for LTBI and pre defined post treatment time points

SECONDARY OUTCOMES:
Evaluate the immune phenotype and functionality of tissue resident immune cells obtained by bronchoalveolar lavage in subjects with LTBI and either: 1) structural lung damage from prior treated/healed pulmonary tuberculosis or 2) recent prolonge... | Pre Treatment for LTBI and pre defined post treatment time points LTBI and pre definedpost treatment timepoints
Define the role of stable long lasting antigen-specific IL-2 producing CD4+ central memory T cells in identifying subsets of patients with LTBI | Pre Treatment for LTBI and pre defined post treatment time points LTBI and pre defined post treatment timepointspoints

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Nutman, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Montgomery County Public Health Services, TB, Refugee and Migrant Health, Silver Spring, Maryland

REFERENCES:
- [Background] Elias D, Akuffo H, Pawlowski A, Haile M, Schon T, Britton S. Schistosoma mansoni infection reduces the protective efficacy of BCG vaccination against virulent Mycobacterium tuberculosis. Vaccine. 2005 Feb 3;23(11):1326-34. doi: 10.1016/j.vaccine.2004.09.038. PMID 15661380
- [Background] Flynn JL, Chan J. Immunology of tuberculosis. Annu Rev Immunol. 2001;19:93-129. doi: 10.1146/annurev.immunol.19.1.93. PMID 11244032
- [Background] Ewer K, Millington KA, Deeks JJ, Alvarez L, Bryant G, Lalvani A. Dynamic antigen-specific T-cell responses after point-source exposure to Mycobacterium tuberculosis. Am J Respir Crit Care Med. 2006 Oct 1;174(7):831-9. doi: 10.1164/rccm.200511-1783OC. Epub 2006 Jun 23. PMID 16799072